CLINICAL TRIAL: NCT03250871
Title: Hypnosis Contribution to Interventional Electrophysiology Performed Under Local Anesthesia and Morphine Titration Study PAINLESS : Does Hypnosis Reduce Pain in Electrophysiology Procedures ?
Brief Title: Hypnosis in Interventional Electrophysiology
Acronym: PAINLESS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Poitiers University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2017-A01936-47
Record Dates: First submitted 2017-08-11; First posted 2017-08-16 (Actual); Last update posted 2020-02-10 (Actual); Status verified 2019-12

CONDITIONS: Flutter, Atrial; Over 18 Years Old
MeSH Terms: conditions — Atrial Flutter | interventions — Hypnosis

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): Placebo will be the suggestion of self-relaxation methods (for example, "try to relax" ,"try to think of pleasant moment ") and the diffusion of "white noise" during surgery.
  Interventions: Other: Placebo
- Hypnosis (Experimental): Hypnosis will be associated with the usual anesthesia. Hypnosis is a temporary modification of consciousness technique based on suggestion.
  It is divided into three phases:
  * induction: attention of the patient fixed on an object or a part of the body,
  * the dissociation where the patient cuts off auditory, visual and tactile perceptions,
  * and finally the opening towards a hypnotic experience thanks to the imaginary.
  Interventions: Other: Hypnosis

INTERVENTIONS:
Other: Hypnosis — Hypnosis will be supervised by a nurse trained by the French Institute of Hypnosis.
  Arms: Hypnosis
Other: Placebo — Placebo consists in non-hypnotic relaxation suggestions and in hearing white noise through headphones
  Arms: Placebo

SUMMARY:
Hypnosis has already shown to decrease pain and anxiety in different surgical specialities. Nevertheless, its input has never been studied in cardiology. This research is a prospective, monocentric, controlled and randomized study.

Patients over 18 years old and hospitalized for atrial flutter ablation may be included and randomized into one of the arms: placebo or hypnosis.

Global pain will be assessed by a visual analogue pain scale. Anxiety, morphine consumption, and patient sedation will also be assessed.

The aim of this study is to improve the care given to patient undergoing atrial flutter ablation.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Surgery ablation of atrial flutter
* Agreement to participate of the study

Exclusion Criteria:

* Person who does not speak French or deaf
* Chronic pain with the visual analogue scale > 5
* Psychiatric pathology
* Contraindication to paracetamol, lidocaine, morphine
* Pregnant women, or breast-feeding women or without effective contraception

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 116 (Actual)
Dates: Start 2017-10-02 (Actual); Primary Completion 2019-09-23 (Actual); Study Completion 2019-09-26 (Actual)

PRIMARY OUTCOMES:
Global pain self-assessment during the procedure | Collected 45 min after the procedure
  Assessed with visual analogue pain scale

SECONDARY OUTCOMES:
Anxiety during the procedure | Collected after the procedure
  Visual analog scale self-assessment
Morphine consumption | Collected after the procedure
  milligram
Patient sedation evaluation | Collected after the procedure
  numerical rating scale; Externally assessed by the electrophysiologist
Pain assessed prospectively during the procedure; | Evaluated every 5 minutes during the procedure;
  Numerical rating scale score

CONTACTS AND LOCATIONS:
Locations (1):
- CHU DE Poitiers, Poitiers, France